CLINICAL TRIAL: NCT03445637
Title: Post Marketing Surveillance Study to Observe Safety and Efficacy of IBRANCE®
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5481065; NCT03445637 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2018-01-31; First posted 2018-02-26 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Breast Neoplasm
Keywords: Metastatic breast cancer; safety; ibrance
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

SUMMARY:
This non-interventional study is designated as a Post Marketing Surveillance Study and is a commitment to Ministry of Food and Drug Safety (MFDS).

Before the approval of IBRANCE® in Korea, as a part of Risk Management Plan (RMP), which is required by MFDS, safety and efficacy information of new medication will be provided at minimum 1,000 participants administered in the setting of routine practice during the initial 9 years after the approval.

ELIGIBILITY:
Inclusion Criteria

* Women of ≥18 years of age with proven diagnosis of advanced/metastatic breast cancer (locoregionally recurrent or metastatic disease).
* Estrogen Receptor+ (ER+) and/or Progesterone Receptor+ (PgR+) tumor based on local laboratory results (test as per local practice).
* Human Epidermal Growth Factor Receptor 2 -(HER2-) breast cancer based on local laboratory results (test as per local practice or local guidelines)
* Patients must be appropriate candidates for hormone therapy.
* Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study.
* During the post marketing surveillance (PMS) period, patients who initially administer IBRANCE®

Exclusion Criteria

* Known hypersensitivity to letrozole or its excipients or to any Cyclin-Dependent Kinase 4/6 (CDK4/6) inhibitor excipients.
* Pregnant women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: All participants enrolled should meet the usual prescribing criteria for IBRANCE® as per the Local Product Document (LPD) and should be entered into the study at the physician's discretion.
Sampling Method: Probability Sample
Enrollment: 552 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2025-07-13 (Actual); Study Completion 2025-07-13 (Actual)

PRIMARY OUTCOMES:
Treatment-related adverse events during first 3 months | 2018 ~ 2025
  This is a prospective, observational, non-interventional, multi-center study in which subjects will be administered as part of routine practice at Korean health care centers by accredited physicians.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A5481065